CLINICAL TRIAL: NCT06810817
Title: The Effects of Transcranial Direct Current Stimulation and Cognitive Behavioural Programme on Post-stroke Fatigue
Brief Title: Transcranial Direct Current Stimulation and Cognitive Behavioural Programme on Post-stroke Fatigue
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Shamay Ng, Prof, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSEARS20240310002
Record Dates: First submitted 2025-01-28; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation; Physical Conditioning, Human

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- tDCS and cognitive behavioural programme with physical training (Experimental)
  Interventions: Combination Product: tDCS & cognitive behavioral programme with home-based physical training
- sham tDCS and cognitive behavioural programme with physical training (Active Comparator)
  Interventions: Behavioral: sham tDCS & cognitive behavioral programme with home-based physical training
- physical training (Active Comparator)
  Interventions: Behavioral: physical training

INTERVENTIONS:
Combination Product: tDCS & cognitive behavioral programme with home-based physical training — Participants will receive 16 sessions of tDCS and 7 sessions of cognitive behavioral programme over 8 weeks and have physical training at home for 8 weeks.
  Arms: tDCS and cognitive behavioural programme with physical training
Behavioral: sham tDCS & cognitive behavioral programme with home-based physical training — Participants will receive 16 sessions of sham-tDCS and 7 sessions of cognitive behavioral programme over 8 weeks and have physical training at home for 8 weeks.
  Arms: sham tDCS and cognitive behavioural programme with physical training
Behavioral: physical training — Participants will have physical training at home for 8 weeks.
  Arms: physical training

SUMMARY:
This study aims to evaluate the effect of transcranial direct current stimulation and cognitive behavioural programme on fatigue and its related outcomes among people with stroke.

DETAILED DESCRIPTION:
This study will adopt a randomized controlled trial. Participants will be randomized into one of the 3 groups. One group will receive transcranial direct current stimulation and cognitive behavioural programme with home-based physical training. Another group will receive sham transcranial direct current stimulation and cognitive behavioural programme with home-based physical training. One group will receive home-based physical training only.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with stroke at least 6 months ago
* Fatigue Assessment Scale score ≥20
* cognitively intact

Exclusion Criteria:

* Unstable medical conditions leading to fatigue
* Under any clinical trials
* with any other neurological diseases
* history of transient ischemic attack
* Contraindications to tDCS

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Fatigue Assessment Scale | baseline, in the middle during the intervention, immediate post-intervention, 1- and 3-month after the completion of the intervention

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | baseline, in the middle during the intervention, immediate post-intervention, 1- and 3-month after the completion of the intervention
Geriatric Depression Scale | baseline, in the middle during the intervention, immediate post-intervention, 1- and 3-month after the completion of the intervention
Reintegration to Normal Living Index | baseline, in the middle during the intervention, immediate post-intervention, 1- and 3-month after the completion of the intervention
Cardio-ankle vascular index | baseline, in the middle during the intervention, immediate post-intervention, 1- and 3-month after the completion of the intervention
performance fatigue index | baseline, in the middle during the intervention, immediate post-intervention, 1- and 3-month after the completion of the intervention
psychomotor vigilance task | baseline, in the middle during the intervention, immediate post-intervention, 1- and 3-month after the completion of the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No